CLINICAL TRIAL: NCT01521377
Title: A Randomised, Placebo-controlled, Incomplete Block, Four Period Crossover , Repeat Dose Study to Evaluate the Effect of the Inhaled GSK573719/Vilanterol Combination and GSK573719 Monotherapy on Electrocardiographic Parameters, With Moxifloxacin as a Positive Control, in Healthy Subjects.
Brief Title: QTc Study GSK573719+GW642444
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114635
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: LAMA; Respiratory; COPD; Tolerability; Beta-2 Agonist; Safety; Pharmacokinetics; Pharmacodynamics; LABA; Muscarinic Receptor Agonist; Healthy subjects; Moxifloxacin; Anticholinergic; GW642444; GSK573719; QTc
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Moxifloxacin; GSK573719; vilanterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Placebo (Placebo Comparator): Single inhalation from matching placebo dry powder inhaler once daily on days 1-10. Single dose placebo oral tablet moxifloxacin.
  Interventions: Drug: Placebo Moxifloxacin; Drug: Placebo DPI
- Moxifloxacin Positive (Active Comparator): Single inhalation from matching placebo dry powder inhaler once daily on days 1-10. Single dose oral tablet moxifloxacin (400mg) on day 10.
  Interventions: Drug: Moxifloxacin; Drug: Placebo DPI
- GSK573719 Supra-therapeutic dose (Experimental): Single inhalation from GSK573719 (500 microgram) dry powder inhaler once daily on days 1-10. Single dose placebo oral moxifloxacin.
  Interventions: Drug: Placebo Moxifloxacin; Drug: GSK573719
- GSK573719/Vilanterol Therapeutic dose (Experimental): Single inhalation from GSK573719/Vilanterol (125/25 microgram) dry powder inhaler once daily on days 1-10. Single dose placebo oral tablet moxifloxacin on day 10.
  Interventions: Drug: Placebo Moxifloxacin; Drug: GSK573719/Vilanterol 125/25mcg
- GSK573719/Vilanterol Supra-therapeutic dose (Experimental): Single inhalation from GSK573719/Vilanterol (500/100 microgram) dry powder inhaler once daily on days 1-10. Single dose placebo oral tablet moxifloxacin on day 10.
  Interventions: Drug: Placebo Moxifloxacin; Drug: GSK573719/Vilanterol 500/100mcg

INTERVENTIONS:
Drug: Placebo Moxifloxacin — Single dose placebo oral tablet Moxifloxacin
  Arms: GSK573719 Supra-therapeutic dose; GSK573719/Vilanterol Supra-therapeutic dose; GSK573719/Vilanterol Therapeutic dose; Placebo
Drug: Moxifloxacin — Single oral dose tablet Moxifloxacin (400mg)
  Arms: Moxifloxacin Positive
Drug: GSK573719/Vilanterol 125/25mcg — Single inhalation from GSK573719/Vilanterol 125/25mcg DPI once daily
  Arms: GSK573719/Vilanterol Therapeutic dose
Drug: GSK573719 — Single inhalation from GSK573719 500mcg DPI once daily
  Arms: GSK573719 Supra-therapeutic dose
Drug: GSK573719/Vilanterol 500/100mcg — Single inhalation from GSK573719/Vilanterol 500/100mcg DPI once daily
  Arms: GSK573719/Vilanterol Supra-therapeutic dose
Drug: Placebo DPI — Single Inhalation from matching Placebo DPI once daily
  Arms: Moxifloxacin Positive; Placebo

SUMMARY:
This is a randomized, placebo controlled, four period incomplete block,crossover thorough QT study to estimate the effect of repeat dose GSK573719/GW642444M (Vilanterol) combination and GSK573719 monotherapy on the QTc interval in healthy male and female subjects compared with placebo. At least 100 subjects will receive, four of five possible, 10-day repeat dose treatments. Treatments are placebo with a moxifloxacin placebo on day 10, placebo with moxifloxacin (400mg) on day 10, GSK573719/Vilanterol combination (125/25μg) with moxifloxacin placebo on day 10, GSK573719/Vilanterol combinatio (500/100μg) with moxifloxacin placebo on day 10, or GSK573719 (500μg) with a moxifloxacin placebo on day 10. All treatments are double blind except for moxifloxacin (400mg) and moxifloxacin placebo controls, given as a single-blind single dose on Day 10 of the appropriate treatment period.

Primary endpoints are individual time-matched changes from baseline QTcF for GSK573719/Vilanterol combination (125/25μg) and GSK573719 (500μg), 0-24 hours after dosing on Day 10. Secondary endpoints will include individual time-matched changes from baseline in QTcF for GSK573719/Vilanterol combination (500/100μg) and moxifloxacin (400mcg) 0-24 hours after dosing on Day 10. Also changes from baseline in QTci, QTcB, QT, QRS, RR, PR and ventricular rate at each time point after 10 days dosing of each GSK573719 and GSK573719/Vilanterol treatment and single dose moxifloxacin (400mg). Maximal change from baseline 0-24hours after dosing on day 10 will be derived for QTcF, QTci and QTcB for each treatment. Plasma concentrations on Day 10 (0-24 hours) and pharmacokinetic parameters of GSK573719 and Vilanterol will also be derived. Key assessments: 12- lead electrocardiogram (ECG), pharmacokinetics. Safety will be assessed by blood pressure, heart rate, clinical laboratory safety tests and collection of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator believes that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol <40 pg/ml (<147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
  * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until after the Follow Up visit
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Body weight ≥ 45 kg and BMI within the range 18 - 29.5 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* No significant abnormality on 12-lead ECG at screening, including the following specific requirements:

  * Ventricular rate ≥ 40 beats per minute
  * PR interval ≤ 210msec
  * Q waves < 30msec (up to 50 ms permitted in lead III only)
  * QRS interval to be ≥ 60msec and < 120msec
  * The waveforms must enable the QT interval to be clearly defined
  * QTcF interval must be < 450msec (machine or manual reading).
* A 24 hour Holter ECG at screening that demonstrates no clinically significant abnormalities or finding that could interfere with interpretation of the study results, when assessed by an appropriately trained and experienced reviewer
* Subjects who are able to use the Novel DPIsatisfactorily.
* Capable of giving written informed consent and a signed and dated written informed consent is obtained, which includes compliance with the requirements and restrictions listed in the consent form.
* Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked)).
* Available to complete the study.

Exclusion Criteria:

* History or presence of any medically significant disease, or any disorder that would introduce additional risk or interfere with the study procedures or outcome. In particular, a family history of QT prolongation, of early or sudden cardiac death or of early cardiovascular disease.
* History of symptomatic arrhythmias.
* A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHG) at screening.
* A supine mean heart rate outside the range 40-90 beats per minute (BPM) at screening.
* History of tendon disease/disorder related to quinolone treatment.
* History of sensitivity to any of the study medications, including moxifloxacin, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In particular, the subject has a known allergy or hypersensitivity to quinolones, ipratropium bromide, tiotropium, atropine and any of its derivatives. Or any adverse reaction including immediate or delayed hypersensitivity to any β2 agonist or sympathomimetic drug,
* Severe Milk Protein allergy
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

  * an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Consumption of seville oranges, pummelos (members of the grapefruit family) or grapefruit juice from 7 days prior to the first dose of study medication.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 3 month period.
* Pregnant females as determined by positive serum β-HCG test at screening or serum/ urine β-HCG prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Urinary cotinine levels indicative of smoking or history or regular use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12-19 (Actual); Primary Completion 2012-06-05 (Actual); Study Completion 2012-06-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF Interval with GSK573719/ Vilanterol 125/25mcg | Screening, Day 1, and Day 10
  To estimate the effect of GSK573719/ Vilanterol 125/25mcg on the QTcF interval as compared with placebo after 10 days dosing.
Change from baseline in QTcF Interval with GSK573719 500 mcg | Screening, Day 1, and Day 10
  To estimate the effect of GSK573719 500 mcg (four times the highest combination dose being evaluated in Phase III trials) on the QTcF interval as compared with placebo after 10 days dosing.

SECONDARY OUTCOMES:
Change from baseline in QTcF interval with GSK573719/Vilanterol 500/100mcg | Screening, Day 1, and Day 10
  To estimate the effect of GSK573719/ Vilanterol 500/100mcg (four times the highest combination dose being evaluated in Phase III trials) on the QTcF interval as compared with placebo after 10 days dosing.
Change from baseline in QTci and QTcB interval for GSK573719/Vilanterol 125/25mcg and 500/100mcg as compared with timematched placebo. | Screening, Day 1, and Day 10
  To estimate the effect of GSK573719/Vilanterol 125/25mcg and 500/100mcg on the QTci and QTcB interval interval as compared with placebo after 10 days dosing.
Change from baseline in QTci and QTcB interval for GSK573719 500mcg as compared with time-matched placebo. | Screening, Day 1, and Day 10
  To estimate the effect of GSK573719 500mcg, on the QTci and QTcB interval interval as compared with placebo after 10 days dosing.
Change from baseline in QTcF interval for moxifloxacin as compared with time-matched placebo. | Screening, Day 1, and Day 10
  To estimate the effect of a single oral dose of 400mg moxifloxacin on the QTcF interval as compared with placebo on day 10.
Change from baseline in QTci and QTcB interval for moxifloxacin as compared with time-matched placebo. | Screening, Day 1, and Day 10
  To estimate the effect of a single oral dose of 400mg moxifloxacin on the QTci and QTcB interval interval as compared with placebo on day 10.
Change from baseline at each timepoint on Day 10 for other cardiac electrophysiological parameters: QT, QRS, RR, PR and ventricular rate for each active treatment compared with placebo. | Screening, Day 1, and Day 10
  To estimate the effect of all active treatments on other cardiac electrophysiological parameters as compared with placebo after 10 days dosing.
Plasma concentrations of GSK573719 and Vilanterol and derived pharmacokinetic parameters including Cmax, tmax and AUC(0-τ). | Screening, Day 1, and Day 10
  To characterise the pharmacokinetic profiles of GSK573719 and Vilanterol when administered in combination via novel DPI.
Plasma concentrations of GSK573719 and derived pharmacokinetic parameters including Cmax, tmax and AUC(0-τ). | Screening, Day 1, and Day 10
  To characterise the pharmacokinetic profile of supra-therapeutic dose of GSK573719 when administered as monotherapy via novel DPI.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 114635 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114635?search=study&search_terms=114635#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register